CLINICAL TRIAL: NCT06731764
Title: Novel Approaches to the Treatment of Hypothyroidism
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Francesco Celi, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-186-1
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Levothyroxine alone (Active Comparator): Patients in this arm will be administered Levothyroxine/Placebo
  Interventions: Drug: Levothyroxine
- Combination therapy liothyronine once daily (Experimental): Patients in the arm will be administered Levothyroxine/Liothyronine with Liothyronine administered once daily plus placebo
  Interventions: Drug: Levothyroxine; Drug: Levothyroxine/Liothyronine once daily
- Combination therapy liothyronine twice daily (Experimental): Patients in this arm will be administered Levothyroxine/Liothyronine with Liothyronine administered twice daily.
  Interventions: Drug: Levothyroxine; Drug: Levothyroxine/Liothyronine twice daily

INTERVENTIONS:
Drug: Levothyroxine — Patients will receive Levothyroxine/Placebo
  Levothyroxine/Liothyronine with Liothyronine administered twice daily.
  Other Names: LT4
Drug: Levothyroxine/Liothyronine once daily — Patients will receive Levothyroxine/Liothyronine with Liothyronine administered once daily;
  Other Names: LT4/LT3
  Arms: Combination therapy liothyronine once daily
Drug: Levothyroxine/Liothyronine twice daily — Patients will receive Levothyroxine/Liothyronine with Liothyronine administered twice daily;
  Other Names: LT4/LT3
  Arms: Combination therapy liothyronine twice daily

SUMMARY:
Hypothyroidism is a common condition, more frequent in females, associated with excess of cardiovascular risk and poor quality of life not completely abrogated by treatment with levothyroxine.

There is an unmet need to define a safe, effective, and feasible regimen to be applied in large trials aimed at assessing levothyroxine/liothyronine combination therapy in patients living with hypothyroidism.

To address this knowledge gap we propose a randomized, three-arm, double-blind, controlled, escalating dose parallel pilot study whose results will lay the foundation of large multicenter trial(s) able to demonstrate the effectiveness (or lack thereof) of levothyroxine/liothyronine combination therapy.

DETAILED DESCRIPTION:
Hypothyroidism is a common condition associated with excess of cardiovascular risk and poor quality of life which are not completely abrogated by treatment with levothyroxine (synthetic T4, LT4), potentially because of the inability to compensate for the loss of T3 secreted by the thyroid gland. Experimental data in animal models indicate that only combination LT4 and liothyronine (synthetic T3, LT3) can restore normal concentrations of thyroid hormones across the tissues target of the hormonal action. Clinical trials based on LT4/LT3 combination therapy and desiccated thyroid extracts (containing T3) have provided conflicting data, but the plurality of the results indicates a preference toward T3-containing therapies when compared to LT4 alone. Conversely, the short half-life of T3 poses concern of cardiovascular toxicity due to fluctuating levels of T3, particularly when LT3 is prescribed in single dose. No study has systematically assessed the optimal dose and frequency of LT3 administration in LT4/LT3 combination therapy. There is an unmet need to define a safe, effective, and feasible regimen to be applied in large trials aimed at assessing LT4/LT3 therapy efficacy and safety.

We have conducted clinical studies aimed at characterizing the pharmacokinetics and pharmacodynamics of LT3 and, more recently, we completed a R21-sponsored LT4/LT3 combination therapy clinical trial in patients undergoing total thyroidectomy. The data suggest that LT4/LT3 combination therapy is effective in normalizing thyroid hormone levels and in preventing the rise in serum cholesterol and weight when compared to LT4 alone. Moreover, our results from a prior study appear to negate a clinical role of rapid T3 action, supporting the use of LT3 in single administration. These original findings serve as foundation for the current proposal.

Hypothesis: A once daily administration of LT4/LT3 combination therapy will be (i) effective yet safe, (ii) comparable to a twice daily LT4/LT3 administration regimen, and (iii) superior to LT4 therapy in improving clinically relevant indices of thyroid hormone action.

To test this hypothesis, we propose a randomized, three-arm, double-blind, controlled, escalating dose parallel pilot study in which 90 patients with hypothyroidism (30 each group) will be randomized to six months of treatment with LT4, LT4/LT3 with LT3 once daily, or LT4/LT3 with LT3 twice daily.

This novel and rigorous study based on our original observations will fill the knowledge gap of effects and dosing of LT4/LT3 combination therapy, laying the foundation for large multicenter trial(s) able to demonstrate the effectiveness (or lack thereof) of LT4/LT3 combination therapy, fulfilling the aims of PAS-23-086.

ELIGIBILITY:
Inclusion Criteria:

History of hypothyroidism Treatment with levothyroxine Levothyroxine dose >1.2 mcg/kg

Exclusion Criteria:

Body weight <50 or >100 Kg.

Indication for TSH suppression (high risk follicular-derived thyroid cancer).

Secondary (pituitary) hypothyroidism (ICD-10 E23.0); Pregnancy; breastfeeding; uncontrolled diabetes (HbA1c >8.5% at screening); use of oral Semaglutide (Rybelsus); Uncontrolled Hypertension (BP > 140/90 at screening); current use of T3-containing therapies (Liothyronine, desiccated thyroid extracts).

Patients receiving lipid-lowering therapies must maintain the same dose throughout the participation in the study. Changes in lipid lowering therapy/dose will result in termination from the study.

Patients receiving anti-acid (H2 blockers, proton pump inhibitors) therapies must maintain the same dose throughout the participation in the study. Changes in anti-acid therapy/dose will result in termination from the study. Use of other medications known to interfere with the absorption of thyroid hormone, or affecting the thyroid hormone axis (Burch 2019) will be considered exclusion criteria.

Bariatric surgery, initiation of GLP-1 agonist therapy (irrespective of the indication), enrollment in structured weight loss programs will result in dismissal from the study.

Current pregnancy, pregnancy planned within the next 6 months, and lack of contraception in women of reproductive age will be exclusionary. We will verify that the participant is not pregnant through a urine pregnancy test at the time of the first study visit and at each of the follow-up visits. Any participants who become pregnant will terminate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Total Cholesterol | 6 month
  Changes between groups
Changes in LDL Cholesterol | 6 month
  Changes between groups

SECONDARY OUTCOMES:
Changes in Weight | 6 month
  Changes between groups

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Celi, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No